CLINICAL TRIAL: NCT00917852
Title: Evaluation of the GORE Conformable TAG® Thoracic Endoprosthesis for Treatment of Traumatic Transection of the Descending Thoracic Aorta
Brief Title: Evaluation of the GORE Conformable TAG® for Treatment of Traumatic Transection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAG 08-02
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Thoracic Injuries
Keywords: aorta; trauma; transection
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE Conformable TAG® Thoracic Endoprosthesis (Experimental)
  Interventions: Device: Gore Conformable TAG Thoracic Endoprosthesis

INTERVENTIONS:
Device: Gore Conformable TAG Thoracic Endoprosthesis — Endovascular stent graft

SUMMARY:
TAG 08-02 is a prospective, multicenter, single-arm study to evaluate the use of the CTAG Device in traumatic transection of the descending thoracic aorta.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic transection of the DTA that requires repair, determined by the treating physician
2. Traumatic aortic transection location between, but does not include, the left subclavian artery and celiac artery
3. Endovascular repair with the GORE Conformable TAG® Device performed less than or = to 14 days after aortic injury
4. Age greater than or equal to 18 years
5. Proximal and distal landing zone length greater than or equal to 2.0 cm. Landing zones must be in native aorta. Landing zone may include left subclavian artery, if necessary
6. All proximal and distal landing zone inner diameters are between 16-42 mm. Diameter assessed by flow lumen and thrombus, if present; calcium excluded
7. Subject capable of complying with study protocol requirements, including follow-up
8. Informed Consent Form signed by subject or legal representative

Exclusion Criteria:

1. Differing proximal and distal neck diameters (aortic taper) outside the intended aortic diameter requirements (sizing guide) for a single endoprosthesis diameter and the inability to use devices of different diameters (in adherence to the sizing guide) to compensate for the taper
2. Tortuous or stenotic iliac and/or femoral arteries and inability to use a conduit for vascular access
3. Aneurysmal, dissected, heavily calcified, or heavily thrombosed landing zone(s)
4. Infected aorta
5. Subject has a systemic infection and may be at increased risk of endovascular graft infection
6. Planned coverage of left carotid or celiac arteries with the CTAG Device
7. Known degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome
8. Treatment in another drug or medical device study within 1 year of study enrollment
9. Known history of drug abuse
10. Pregnant female
11. Moribund patient not expected to live 24 hours with or without operation, determined by the treating physician
12. Injury Severity Score of 75
13. Subject has known sensitivities or allergies to the device materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Farber, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (26):
- United States (26):
  - Los Angeles, California
  - Stanford, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Lake Success, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Temple, Texas
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Panthofer AM, Olson SL, Harris DG, Matsumura JS. Derivation and validation of thoracic sarcopenia assessment in patients undergoing thoracic endovascular aortic repair. J Vasc Surg. 2019 May;69(5):1379-1386. doi: 10.1016/j.jvs.2018.08.180. Epub 2018 Dec 28. PMID 30598352

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Started | 51
Completed | 45
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Time Frame: 30 days post-treatment
Population: All enrolled subjects
Measure: Number; unit: participants
Arm/Group | GORE Conformable TAG® Device Surgical Implant
Number analyzed (Participants) | 51
participants | 4

2. Primary Outcome: Major Device Events
Description: Major device events requiring reintervention through 1 month study window. Possible device events include but are not limited to endoleak, migration, wire fracture, compression, erosion, extrusion, aortic dilatation, endograft infection, and aortic rupture.
Time Frame: 1 month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GORE Conformable TAG® Thoracic Endoprosthesis
Number analyzed (Participants) | 51
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | CTAG Device Trauma Subjects
All-Cause Mortality (participants affected / at risk) | 7/51
Serious Adverse Events (participants affected / at risk) | 27/51
Other Adverse Events (participants affected / at risk) | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTAG Device Trauma Subjects (N=51)
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Complication associated with device (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fat embolism (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1
Splenic injury (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Blood culture positive (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral hypoperfusion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hyponatraemic seizure (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haemodynamic instability (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Intermittent claudication (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTAG Device Trauma Subjects (N=51)
Anaemia (Blood and lymphatic system disorders) | 10
Leukocytosis (Blood and lymphatic system disorders) | 3
Angina pectoris (Cardiac disorders) | 8
Atrial fibrillation (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 9
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 4
Generalised oedema (General disorders) | 3
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 10
Pneumonia (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 5
Mental status changes (Psychiatric disorders) | 3
Post-traumatic stress disorder (Psychiatric disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6
Deep vein thrombosis (Vascular disorders) | 3
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.